CLINICAL TRIAL: NCT04504539
Title: Comparison of mOPV1 Schedules for Routine Immunization in Pakistan. A Community Based Randomized Control Trial
Brief Title: Use of mOPV1 in Routine Immunization in Pakistan.
Acronym: mOPV1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Ali Faisal Saleem, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-3284-11191
Record Dates: First submitted 2020-07-23; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Oral Polio Vaccine
Keywords: mOPV; bOPV; randomized trial

STUDY DESIGN:
Intervention Model Description: Different regimens of mOPV and bOPV in combination with either fractional IPV (fIPV) or full dose IPV (FIPV) will be used.
Who Masked: Participant, Outcomes Assessor
Masking Description: The mOPV and bOPV vaccine vials will be masked by the Clinical Trials Unit to look identical. The assessor will only be provided the enrollment ID and will not be aware of the participant's randomization status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mOPV with FIPV (Experimental): mOPV vaccine will be given at birth, 6 weeks, 10 weeks and 14 weeks of age along with a single dose of FIPV at 14 weeks of age.
  Interventions: Biological: mOPV; Biological: Full dose IPV; Biological: fractional IPV
- bOPV with FIPV (Experimental): bOPV vaccine will be given at birth, 6 weeks, 10 weeks and 14 weeks of age along with a single dose of FIPV at 14 weeks of age.
  Interventions: Biological: bOPV; Biological: Full dose IPV; Biological: fractional IPV
- mOPV with fIPV (Experimental): mOPV vaccine will be given at birth, 6 weeks, 10 weeks and 14 weeks of age along with a two doses of fIPV at 6 weeks and 14 weeks of age.
  Interventions: Biological: mOPV; Biological: Full dose IPV; Biological: fractional IPV
- bOPV with fIPV (Experimental): bOPV vaccine will be given at birth, 6 weeks, 10 weeks and 14 weeks of age along with a two doses of fIPV at 6 weeks and 14 weeks of age.
  Interventions: Biological: bOPV; Biological: Full dose IPV; Biological: fractional IPV

INTERVENTIONS:
Biological: mOPV — mOPV (monovalent oral polio vaccine) is an oral polio vaccines which consists of only attenuated virus of serotypes 1
  Arms: mOPV with FIPV; mOPV with fIPV
Biological: bOPV — bOPV (bivalent oral polio vaccine) is an oral polio vaccines which consists of attenuated virus of serotypes 1and 3
  Arms: bOPV with FIPV; bOPV with fIPV
Biological: Full dose IPV — FIPV (full dose injectable polio vaccine)
Biological: fractional IPV — fIPV (fractional dose injectable polio vaccine)

SUMMARY:
Pakistan has uninterrupted circulation of polioviruses and this may threaten the entire global community. Bivalent OPV (bOPV), which protects against types 1 and 3, is used for routine immunization. However, type-3 wild poliovirus is on the verge of eradication, therefore mOPV1 is important to achieve eradication of type-1 poliovirus.

The main rationale of the study is to interrupt WPV1 circulation and stopping the outbreaks of VDPVs with the help of mOPV1 instead of bOPV2 for routine immunization, which contains live poliovirus, and will eventually lead to complete eradication and containment of type 1 WPV, vaccine-related (VDPV) and Sabin polioviruses. This study will provide data to National Immunization Authorities in order to make strategic decisions about their polio vaccination schedules in anticipation of the potential global bOPV2 to mOPV1 switch and will provide data on the proposed responses to type 1 poliovirus outbreaks.

DETAILED DESCRIPTION:
Wild Polio Virus 1 (WPV1) is the only responsible virus for wild polio cases across the globe. The world has successfully eradicated wild poliovirus (PV) 2 and 3. Poliomyelitis eradication has entered its last phase with only three remaining endemic countries, of which Pakistan is one and has highest number of WPV1 cases in 2019. The main stream strategies by the Global Polio Eradication Initiative has made the substantial progress towards the eradication of poliomyelitis ever since the World Health Assembly has sanctioned it as an emerging global Public Health threat. These strategies focus on high-quality immunization activities (routine and supplemental) that target children from birth to age 5 years with oral poliovirus vaccines (OPVs), and maintaining a system for acute flaccid paralysis surveillance.

Pakistan has uninterrupted circulation of polioviruses and this may threaten the entire global community and implies impending failure of goal of global eradication. According to the Polio endgame strategy 2019-2023, Pakistan and Afghanistan are the only countries in which WPV transmissions continues to be reported. The genetic sampling and environmental surveillance have revealed that WPV1 has predominantly persisted in Pakistan and Afghanistan and are closely linked as they constitute one epidemiological block. Bivalent OPV (bOPV), which protect against types 1 and 3, is used for routine immunization. However, type-3 wild poliovirus is on the verge of eradication, therefore mOPV1 is important to achieve eradication of type-1 poliovirus whose appearance has been continually been confirmed by the genetic and environmental samplings.

The main rationale of the study is to interrupt WPV1 circulation and stopping the outbreaks of VDPVs with the help of mOPV1 instead of bOPV2 for routine immunization, which contains live poliovirus, and will eventually lead to complete eradication and containment of type 1 WPV, vaccine-related (VDPV) and Sabin polioviruses. The study rationale is in line with the Goal 1- Eradication of GPEI. This study will provide data to National Immunization Authorities in order to make strategic decisions about their polio vaccination schedules in anticipation of the potential global bOPV2 to mOPV1 switch and will provide data on the proposed responses to type 1 poliovirus outbreaks.

Research Questions and Main Objectives :

Overall Objectives of the study will be:

* To assess the serum immunity against type 1,2 and 3 polioviruses achieved with two different mOPV1 routine immunization schedule (mOPV1+fIPV (fractional dose intradermal IPV); mOPV1+FIPV (full dose intramuscular IPV))
* To compare the serum immunity against type 1,2 and 3 polioviruses achieved with two different mOPV1 routine immunization schedule with bOPV2 routine immunization schedules (mOPV1+fIPV, mOPV1+FIPV with bOPV2+fIPV, bOPV2+FIPV)
* To assess the type 2 response after One full dose IPV with mOPV1 and bOPV2 routine immunization schedule
* To assess the type 2 response after two fractional doses of IPV with mOPV1 and bOPV2 routine immunization schedule

ELIGIBILITY:
Inclusion Criteria:

* born healthy with birth weight 2.0 kg or more, with immediate cry.

  * Parents resident of the study areas Not planning to travel away during entire the study period (birth-154 days; birth - 22 weeks) for 3 months at the time of enrolment
  * Parent/guardian provides informed consent

Exclusion Criteria:

* Refusal of blood testing and cord blood testing

  * Receipt of OPV after birth before eligibility screen
  * Newborns with certain medical conditions i.e., syndromic infants, neonate with petechial or purpura (contraindication of intramuscular injections)
  * A confirmed diagnosis of immunodeficiency disorder in a blood relative will render the newborn ineligible for the study.

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 560 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of children with change in antibody titres following vaccination | This will be checked in samples taken at birth, 6 weeks post vaccination, 10 weeks, 14 weeks and 18 weeks of age
  The number of children who produce antibodies following vaccination of each of the 4 arms

CONTACTS AND LOCATIONS:
Overall Officials: Ali Saleem, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No